CLINICAL TRIAL: NCT00005896
Title: Phase I Pilot Study of CD34 Enriched, Fanconi's Anemia Complementation Group C Gene Transduced Autologous Peripheral Blood Stem Cell Transplantation in Patients With Fanconi's Anemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Minnesota (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/15107; UMN-MT-1997-10; UNM-MT-9710
Record Dates: First submitted 2000-06-02; First posted 2000-06-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-03

CONDITIONS: Fanconi's Anemia
Keywords: Fanconi's anemia; aplastic anemia; hematologic disorders; rare disease
MeSH Terms: conditions — Fanconi Anemia; Anemia, Aplastic; Hematologic Diseases; Rare Diseases | interventions — Filgrastim

INTERVENTIONS:
Drug: filgrastim
Genetic: Autologous stem cells transduced with FACC retroviral vector
Procedure: Autologous Stem Cell Transplantation

SUMMARY:
OBJECTIVES: I. Determine the safety of transferring the Fanconi anemia complementation group C (FACC) gene to hematopoietic progenitors by retroviral mediated gene transfer in patients with Fanconi's anemia, complementation group C.

II. Determine the extent of engraftment following this treatment regimen without prior ablation of recipient marrow in these patients.

III. Determine the ability of this treatment regimen to correct the cell phenotype and improve hematopoietic function in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive filgrastim (G-CSF) subcutaneously daily on days 0-6 followed by apheresis to collect peripheral blood stem cells (PBSC) on days 5-7. PBSCs are processed in vitro for enrichment of CD34 cells and transduced with a Fanconi's anemia complementation C (FACC) retroviral vector on days 5-10. Patients receive transduced PBSCs IV over no more than 2 hours on days 8-10. PBSC infusions may be repeated no more than every 2 months for up to 4 courses total.

Patients are followed monthly for 3 months, every 3 months for 9 months, every 6 months for the next year, and then yearly thereafter.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Fanconi's anemia, complementation group C (FACC) Confirmed by diepoxybutane or mitomycin testing AND DNA analysis indicating FACC mutations
* Patients at least 25 kg weight
* No acute leukemia OR Bone marrow aspirate with greater than 10% blasts
* No patients who elect bone marrow transplantation

--Prior/Concurrent Therapy--

* At least 14 days since prior therapy for any acute viral, bacterial, or fungal infection

--Patient Characteristics--

* Performance status: Karnofsky 40-100%
* Hepatic: SGOT, SGPT, and alkaline phosphatase no greater than 5 times upper limit of normal (ULN) PT/PTT no greater than 1.5 times ULN Serum amylase no greater than 1.5 times ULN Bilirubin no greater than 2.5 mg/dL Triglyceride less than 400 mg/dL
* Renal: Creatinine clearance greater than 50 mL/min
* Cardiovascular: Normal cardiac function No ischemic heart disease that may be considered an anesthetic or operative risk
* Pulmonary: No lung disease that may be considered an anesthetic or operative risk Resting transcutaneous oxygen saturation greater than 90% on room air
* Other: HIV negative Hepatitis B surface antigen negative No underlying condition that may preclude study therapy (e.g., allergies to study reagents)
* No acute viral, bacterial, or fungal infection Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6
Dates: Start 2000-03

CONTACTS AND LOCATIONS:
Overall Officials: John E. Wagner, Jr., Study Chair — Masonic Cancer Center, University of Minnesota